CLINICAL TRIAL: NCT01149473
Title: A Relative Bioavailability Study of Losartan Potassium/Hydrochlorothiazide 100/25 mg Tablets Under Non-Fasting Conditions
Brief Title: Losartan Potassium/Hydrochlorothiazide 100/25 mg Tablets in Healthy Subjects Under Non-Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Responsible Party: Associate Director, Biopharmaceutics, Teva Pharmaceuticals USA
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: B046515
Record Dates: First submitted 2010-06-21; First posted 2010-06-23 (Estimated); Results first posted 2010-09-14 (Estimated); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — hydrochlorothiazide, losartan drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Generic Test Product (Experimental): Losartan potassium/Hydrochlorothiazide 100/25 mg Tablets
  Interventions: Drug: Losartan potassium/Hydrochlorothiazide
- Reference Listed Drug (Active Comparator): Hyzaar® 100/25 mg Tablets
  Interventions: Drug: Losartan potassium/Hydrochlorothiazide

INTERVENTIONS:
Drug: Losartan potassium/Hydrochlorothiazide — 100/25 mg Tablets
  Arms: Generic Test Product
Drug: Losartan potassium/Hydrochlorothiazide — 100/25 mg Tablets
  Other Names: Hyzaar®
  Arms: Reference Listed Drug

SUMMARY:
The objective of this study is to compare the relative bioavailability of Losartan potassium/Hydrochlorothiazide 100/25 mg tablets (manufactured by Teva Pharmaceutical Industries, Ltd. and distributed by Teva Pharmaceuticals USA) with that of Hyzaar® 100/25 mg tablets (Merck) in healthy, adult, non-smoking subjects under non-fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA Bioequivalence Statistical Methods

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking, male and female subjects at least 18 years of age.
* BMI (body mass index) of 30 or less.
* Females in this study must be physically unable to become pregnant (postmenopausal for at least 6 months or surgically sterile).
* Successful completion of a physical examination within 28 days of initiation of the study.
* Negative serum pregnancy test (females).

Exclusion Criteria:

* Subjects with a significant recent history of chronic alcohol consumption (past 2 years), drug addiction, or serious gastrointestinal, renal, hepatic, or cardiovascular disease, tuberculosis, epilepsy, asthma (past 5 years), diabetes, psychosis, or glaucoma will not be eligible for this study.
* Subjects whose clinical laboratory test values are outside the reference range and are deemed clinically significant by the Principle Investigator.
* Subjects who have a history of allergic responses to the classes of drugs being tested will be excluded from the study.
* Subjects who use tobacco in any form will not be eligible to participate in the study. 3 months abstinence is required.
* Subjects found to have urine concentrations of any of the tested drugs of abuse will not be allowed to participate.
* Subjects should not have donated blood and/or plasma for at least 30 days prior to the first dosing of the study.
* Subjects who have taken any investigational drug within 30 days prior to the first dosing of the study will not be allowed to participate.
* Female subjects who are pregnant or who are able (women with child bearing potential) to become pregnant during the study will not be allowed to participate.
* All female subjects will be screened for pregnancy at check-in each study period. Subjects with positive or inconclusive results will be withdrawn from the study.
* Subjects who do not tolerate venipuncture will not be allowed to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2004-03; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D Carlson, Pharm D, Principal Investigator — PRACS Institute, Ltd.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Losartan/HCTZ (Test) First: 100/25 mg Losartan potassium/Hydrochlorothiazide test product dosed in first period followed by 100/25 mg Hyzaar® Tablets reference product dosed in the second period.
- Hyzaar® (Reference) First: 100/25 mg Hyzaar® Tablets reference product dosed in first period followed by 100/25 mg Losartan potassium/Hydrochlorothiazide test product dosed in the second period.
Period: First Intervention
Arm/Group | Losartan/HCTZ (Test) First | Hyzaar® (Reference) First
Started | 40 | 40
Completed | 39 | 39
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1
Period: Washout of 7 Days
Arm/Group | Losartan/HCTZ (Test) First | Hyzaar® (Reference) First
Started | 39 | 39
Completed | 38 | 38
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Second Intervention
Arm/Group | Losartan/HCTZ (Test) First | Hyzaar® (Reference) First
Started | 38 | 38
Completed | 38 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Losartan/HCTZ (Test) First | Hyzaar® (Reference) First | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 39 | 79
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 33 | 33 | 66
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 2 | 3
  Black | 3 | 2 | 5
  Caucasian | 35 | 36 | 71
  Hispanic | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Losartan(Maximum Observed Concentration of Drug Substance in Plasma)
Description: Bioequivalence based on Losartan Cmax.
Time Frame: Blood samples collected over a 48 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Losartan/HCTZ (Test): 100/25 mg Losartan potassium/Hydrochlorothiazide test product dosed in either period.
- Hyzaar® (Reference): 100/25 mg Hyzaar® Tablets reference product dosed in either period.
Arm/Group | Losartan/HCTZ (Test) | Hyzaar® (Reference)
Number analyzed (Participants) | 76 | 76
ng/mL | 458.29 (323.345) | 409.324 (251.876)
Statistical Analysis 1: Comparison: Losartan/HCTZ (Test) vs Hyzaar® (Reference); Test type: Non-Inferiority or Equivalence — ANOVA is to be used to identify the source contributions by factors including subjects, period, formulation and potential interactions. The geometric mean ratio together with the ANOVA residual mean error term are used to identify the statistical basis for the 90% confidence interval for the ratio of the population means (Test [T]/Reference[R]) of the identified metrics (e.g. AUC, Cmax); Ratio of the T/R geometric mean x 100 = 109, 90% CI 2-sided [98.1 to 120] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the reference (R) and test (T) product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t of Losartan(Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Bioequivalence based on Losartan AUC0-t.
Time Frame: Blood samples collected over a 48 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Losartan/HCTZ (Test) | Hyzaar® (Reference)
Number analyzed (Participants) | 76 | 76
ng*h/mL | 959.41 (480.988) | 939.492 (465.001)
Statistical Analysis 1: Comparison: Losartan/HCTZ (Test) vs Hyzaar® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 102, 90% CI 2-sided [98.8 to 106] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC0-inf of Losartan(Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Bioequivalence based on Losartan AUC0-inf.
Time Frame: Blood samples collected over a 48 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Losartan/HCTZ (Test) | Hyzaar® (Reference)
Number analyzed (Participants) | 76 | 76
ng*h/mL | 957.445 (465.781) | 956.046 (467.567)
Statistical Analysis 1: Comparison: Losartan/HCTZ (Test) vs Hyzaar® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 101, 90% CI 2-sided [98.6 to 104] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Cmax of Hydrochlorothiazide(Maximum Observed Concentration of Drug Substance in Plasma)
Description: Bioequivalence based on Hydrochlorothiazide Cmax.
Time Frame: Blood samples collected over a 48 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Losartan/HCTZ (Test) | Hyzaar® (Reference)
Number analyzed (Participants) | 76 | 76
ng/mL | 136.361 (33.311) | 132.717 (35.468)
Statistical Analysis 1: Comparison: Losartan/HCTZ (Test) vs Hyzaar® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 103, 90% CI 2-sided [98.8 to 108] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: AUC0-t of Hydrochlorothiazide(Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Bioequivalence based on Hydrochlorothiazide AUC0-t.
Time Frame: Blood samples collected over a 48 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Losartan/HCTZ (Test) | Hyzaar® (Reference)
Number analyzed (Participants) | 76 | 76
ng*h/mL | 917.034 (212.109) | 919.631 (210.684)
Statistical Analysis 1: Comparison: Losartan/HCTZ (Test) vs Hyzaar® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 99.7, 95% CI 2-sided [98.6 to 101] — [estimate comment as in outcome 1, analysis 1]

6. Primary Outcome: AUC0-inf of Hydrochlorothiazide(Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Bioequivalence based on Hydrochlorothiazide AUC0-inf.
Time Frame: Blood samples collected over a 48 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Losartan/HCTZ (Test) | Hyzaar® (Reference)
Number analyzed (Participants) | 76 | 76
ng*h/mL | 943.22 (217.842) | 945.592 (217.269)
Statistical Analysis 1: Comparison: Losartan/HCTZ (Test) vs Hyzaar® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 99.7, 90% CI 2-sided [98.7 to 101] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the study, which was approximately 2 weeks in duration.
Description: Volunteers were monitored throughout the study for any adverse experiences. AEs were collected through both solicited and unsolicited methods. The volunteers were encouraged to report signs, symptoms, and any changes in health to the clinic staff.
Arm/Group | Losartan/HCTZ (Test) | Hyzaar® (Reference)
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 0/80 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.